CLINICAL TRIAL: NCT05486988
Title: A Prospective，Randomized, Multi-center Study to Identify the Patients Who Benefit From Short-course Chemotherapy (2 Cycles) in Combination With Immunotherapy as Treatment for Patients With Locally Advanced Unresectable or Metastatic Non-small Cell Lung Cancer (TLUNG)
Brief Title: ctDNA as a Biomarker for Treatment in Advanced NSCLC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SCOG006
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Circulating Tumor DNA; immunotherapy; chemotherapy (2/4~6 cycles)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immunotherapy; Antineoplastic Agents; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — circulating tumor DNA (ctDNA) of peripheral blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2 cycles chemotherapy combined with PD-1/PD-L1 inhibitors: Participants receive 2 cycles chemotherapy combined with PD-1/PD-L1 inhibitors, after achieving CR/PR/SD according to RECIST v1.1, then will continue immune monotherapy maintenance therapy.
  Interventions: Drug: Immunotherapy; Drug: Chemotherapeutic Agent
- 4-6 cycles chemotherapy combined with PD-1/PD-L1 inhibitors: Participants receive 4~6 cycles chemotherapy combined with PD-1/PD-L1 inhibitors, after achieving CR/PR/SD according to RECIST v1.1, then will continue immune monotherapy maintenance therapy.
  Interventions: Drug: Immunotherapy; Drug: Chemotherapy

INTERVENTIONS:
Drug: Immunotherapy — PD-1/PD-L1 inhibitors
Drug: Chemotherapeutic Agent — 2 cycles
  Groups: 2 cycles chemotherapy combined with PD-1/PD-L1 inhibitors
Drug: Chemotherapy — 4~6 cycles
  Groups: 4-6 cycles chemotherapy combined with PD-1/PD-L1 inhibitors

SUMMARY:
The dynamic monitoring of circulating tumor DNA aims to evaluate the response and progression-free survival of short-course chemotherapy (2 cycles) combined with immunotherapy in patients with locally advanced unresectable or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
For patients with locally advanced unresectable or metastatic non-small cell lung cancers, 4-6 cycles of chemotherapy plus immunotherapy with immune maintenance therapy is currently the standard treatment. Short-course chemotherapy (2 cycles) combined with immunotherapy has been proved effective in some patients. Recently, circulating tumor DNA (ctDNA) has been detected in the cell-free component of peripheral blood samples in advanced non-small cell lung cancers and many other solid tumors. To identify the patients who can benefit from the short-course chemotherapy (2 cycles) combined with immunotherapy, dynamic monitoring of ctDNA in both 4-6 cycles and 2 cycles chemotherapy patients could be a promising alternative test.

ELIGIBILITY:
Inclusion Criteria:

* (1)Histologically confirmed non-small cell lung cancer; (2)Locally advanced unresectable or metastatic disease; (3)Male or female aged over 18 years and under 80 years; (4)Subjects must not have received any immunotherapy for advanced lung cancer, and have an estimated life expectancy of more than 12 weeks (5)Eastern Cooperative Oncology Group (ECOG) score as 0 ~ 1; (6)No EGFR mutation, ALK or ROS1 rearrangement; (7)Adequate tumor tissue for PD-L1 testing; (8)With at least one measurable lesion confirmed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1)； (9)The subjects must sign the informed consent, indicating that they understand the purpose of the study, understand the necessary procedures of the study, and are willing to participate in the study.

Exclusion Criteria:

* (1)Serious immune-related adverse events occurred; (2)Participation in other clinical study; (3)With the history of autoimmune disease or immunodeficiency disease; (4)History of another primary malignancy within 5 years; (5)Without complete clinical information; (6)Pregnant or lactating women; (7)Other conditions in which the investigator believes that the patient should not participate in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female aged over 18 years and under 80 years with locally advanced unresectable or metastatic non-small cell lung cancer, and no prior immunotherapy.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-07-31 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in ctDNA Level Following Chemo-immunotherapy | up to 1 year
  Will be assessed for ctDNA levels at baseline, end of chemotherapy, and immunotherapy maintenance

SECONDARY OUTCOMES:
Progression-free survival | up to 1 year
  From the date of treatment until the date of progression of lung cancer or death from any other cause assessed up to 12 months
Overall survival | up to 24 months
  From the date of treatment until the date of death from any cause assessed up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- 900TH Hospital of Joint Logisti'cs Support Force, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No